CLINICAL TRIAL: NCT06706284
Title: Glycemic and Weight Loss Effects of GLP-1R Agonist Therapy in Subjects With Spinal Cord Injury and Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marzieh Salehi (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Marzieh Salehi, Professor, Division of Diabetes/ Medicine, University of Texas Health Science Center at San Antonio, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000591; R01DK140144-02 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Type 2 Diabetes
Keywords: Glucose regulation; Semaglutide; Ozempic; Glucagon- Like Peptide 1 (GLP-1)
MeSH Terms: conditions — Spinal Cord Injuries; Diabetes Mellitus, Type 2 | interventions — semaglutide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Controlled 2 arm assignment study. The investigators will stochastically match the patient characteristics between the two arms using for a 2:1 design in terms of level of gender (male, female), level of injury (tetraplegia, paraplegia), dichotomized baseline HbA1c (above or below 7.5%), dichotomized age (above or below a median age for this population) and dichotomized BMI (above or below a median BMI for this population)
Who Masked: Participant
Masking Description: Patients will be blinded to the treatment assignment. The study team will be unblinded. The investigators will deliver the treatment assignments to the hospital pharmacist as they occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCI and T2DM Treatment Group (Experimental): Participants with spinal cord injury (SCI) and type 2 diabetes (T2DM) will be assigned to semaglutide weekly for 24 weeks. Semaglutide administration: once-weekly self-administration of SGT, titrated to a dose of 2 mg/week as per FDA approved guidelines. All subjects will be instructed how to inject and titrate up the dose.
  Interventions: Drug: Semaglutide Injectable Product
- SCI and T2DM Placebo Group (Placebo Comparator): Participants with spinal cord injury (SCI) and type 2 diabetes (T2DM) will be assigned to the placebo group and inject normal saline weekly for 24 weeks. All subjects in the placebo group will be instructed how to inject and titrate up the dose to mimic the semaglutide administration to a maximum dose of 2 mg in 12 weeks and then continue for remainder of study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide Injectable Product — A GLP-1 inhibitor used to control T2DM
  Other Names: Ozempic
  Arms: SCI and T2DM Treatment Group
Other: Placebo — Saline solution will be administered with the same frequency as semaglutide and participants will be instructed how to use the saline in the same manner as the active drug group.
  Other Names: Saline solution
  Arms: SCI and T2DM Placebo Group

SUMMARY:
It is not known whether a new diabetes drug, semaglutide, is an effective treatment for type 2 diabetes for persons with spinal cord injury (SCI), a population at higher risk for this condition. Therefore, this study looks at the effect of semaglutide on glucose levels in the body and other information about type 2 diabetes and obesity.

DETAILED DESCRIPTION:
This study consists of 7-9 in-person visits and 9-10 phone visits, and participants will be randomized to either semaglutide or placebo for 24 weeks. The participants first visit, will include review of medical history and performance of standard tests to check the participant's health and eligibility for the study. Before starting any medication, participants will have 2 more visits:

* a mixed meal tolerance test, to examine their body's response to nutrient ingestion and
* a glucose clamp study to examine insulin sensitivity. These tests will be scheduled on two separate days. Following the 3 baseline visits, participants will be randomized to either the intervention (once-weekly injection of semaglutide, also known as Ozempic, for 24 weeks) or placebo. During the 24-week intervention participants will receive 9-10 phone calls to discuss their progress and experiences with the interventions and will also be asked to return for a short research visit including interim medical history with or without blood sample collection twice. At the end of 24 weeks, the treatments will be discontinued, and participants will repeat the meal and glucose studies scheduled over two separate days. During participation, fat/lean mass will be measured using DEXA and liver fat mass may be measured using fibroscan. In addition, participants may be asked for a stool sample.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-70 years (inclusive) at screening
2. More than one year after spinal cord injury
3. Levels if injury C2-L2 with Asia Impairment Scale A, B, C or D.
4. Provision of signed and dated written informed consent prior to any study specific procedures
5. Diagnosed with T2DM with glucose control managed with diet and metformin monotherapy where no significant dose changes (increase or decrease ≥ 50%) have occurred in the three months prior to screening
6. HbA1c 6.0-9.0% at screening
7. BMI > 22 kg/m2 at screening
8. Female subjects of childbearing potential must have a negative pregnancy test at screening and randomization, and must not be lactating
9. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from screening and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study and/or any subject unable or unwilling to follow study procedures.
2. Any subject who has received another investigational product as part of a clinical study within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening
3. Taking mirabegron or other glucose altering medications
4. Taking steroids within the past 1 year
5. Significant anemia (hemoglobin<11g/dL)
6. History of gastric outlet obstruction or chronic diarrhea
7. History of a chronic neurological illness other than SCI (i.e.; MS, etc)
8. Any subject who has received any of the following medications within the specified time-frame prior to the start of the study

   * Herbal preparations or drugs licensed for control of body weight or appetite (eg, orlistat, bupropion-naltrexone, phentermine-topiramate, phentermine, lorcaserin) within a year prior to the start of the study
   * Pioglitazone, SGLT2 or DPPIV inhibitors, GLP-1RA within the last 60 days at the time of screening
9. Severe allergy/hypersensitivity to any of the proposed study treatments, excipients, acetaminophen
10. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus (T1DM) or diabetic ketoacidosis, or if the subject has been treated with daily SC insulin within 90 days prior to screening.
11. Significant inflammatory bowel disease or other severe disease or surgery affecting the upper GI tract (including weight-reducing surgery and procedures) which could affect the interpretation of safety and tolerability data. Prior history of bariatric surgery is not considered exclusion given the ample evidence of safety of use of GLP-1R therapy in this population.
12. Acute or chronic pancreatitis
13. Significant hepatic disease (except for metabolic dysfunction-associated steatohepatitis [MASH] or metabolic dysfunction-associated steatotic liver disease [MASLD]) without portal hypertension or cirrhosis) and/or subjects with any of the following results at screening:

    Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN) Alanine transaminase (ALT) ≥ 3 × ULN Total bilirubin ≥ 2 × ULN
14. Impaired renal function defined as estimated glomerular filtration rate (eGFR) < 45 mL/minute/1.73m2 at screening (GFR estimated according to Modification of Diet in Renal Disease (MDRD) using MDRD Study Equation IDMS-traceable [SI units])
15. Unstable angina pectoris, myocardial infarction, transient ischemic attack (TIA) or stroke within 3 months prior to screening, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
16. Severe congestive heart failure (New York Heart Association Class III or IV)
17. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
18. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer
19. History of HIV infection or other immune compromised disease; and history of organ transplantation
20. Substance dependence or history of alcohol abuse and/or excess alcohol intake
21. Patients on ketogenic diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance | Baseline to 24 weeks
  The change in the incremental AUC Glucose3h response to meal ingestion
Insulin action | Baseline to 24 weeks
  Liver, adipose tissue and muscle insulin sensitivity determined using a two-step euglycemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Salehi, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University Health - Texas Diabetic Institute, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The shared data will be de-identified according to HIPAA and shared under a repository standard Data Use Agreement (DUA).(e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented, as appropriate.ccess to shared data will be controlled according to the repository policy which requires a request and merit review and will be available according to repository processes. The shared data will be de-identified according to HIPAA and shared under a repository standard Data Use Agreement (DUA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be shared as summary results on ClinicalTrials.gov a year after the primary completion date and full results will be shared at study end after data has been analyzed and published in a peer review journal.
Access Criteria: The scientific data generated from this study will be shared in the Texas Digital Library
URL: https://dataverse.tdl.org/